CLINICAL TRIAL: NCT04518423
Title: Prevalence, Determinants and Natural History of Frailty and Pre-frailty in People Over the Age of 65 Years in a Prospective 5-year Observation
Brief Title: Prevalence, Determinants and Natural History of Frailty and Pre-frailty in Elderly People
Acronym: FRAILPOL
Status: Recruiting | Type: Observational
Sponsor: The Opole University of Technology (Other)
Responsible Party: Principal Investigator, Prof Jerzy Sacha, Principal Investigator, The Opole University of Technology
Other Study IDs: FRAILPOL
Record Dates: First submitted 2020-08-12; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Frailty; Frailty Syndrome; Frail Elderly Syndrome; Fragility; Aging; Aging Problems; Aging Disorder; Aging Well
Keywords: Frailty; Physical Frailty; Cognitive Frailty; Social Frailty; Multidimensional Frailty; Elderly; Aging; Frail Scale; Tilburg Frailty Indicator
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly people over the age of 65 years: The study group will comprise community dwelling elderly individuals over the age of 65 years who get around by themselves. The subjects will be followed up for 5 years to investigate the frailty and disability development, and survival.

SUMMARY:
Frailty syndrome (i.e. frailty) is a geriatric syndrome which relies on the reduction of multisystem reserve capacity. Frail people have a lower potential to respond to external stressors and various life incidents as well as they present a weak prognosis particularly in cardiovascular diseases. Yet, frailty is not only a set of physical deficits, but it also concerns psychological and social dimensions of human functioning. Hence, an approach to frailty should be multidimensional because such a concept more adequately reflects a functional degradation in the elderly. Frailty is usually associated with the impaired condition of circulatory system, and therefore, an identification of subclinical cardiovascular abnormalities is paramount in the frailty prevention and treatment. Another potential mechanism which may predispose to frailty is a dysfunction of the autonomic nervous system. This system plays a crucial role in the response to internal or external stressors such as diseases and activities of daily living. An impairment of the autonomic nervous system function may maintain or accelerate the frailty process.

In this scientific project, a comprehensive echocardiography will investigate cardiac function with a particular attention to features which typically change with age, like flow parameters and chambers sizes. The activity of the autonomic nervous system will be explored with the analysis of heart rate, blood pressure and respiratory signals. The study participants will also undergo routine medical examination and a number of additional tests, including: assessment of cognitive function, psychological condition, nutrition status, activities of daily living, and risk of falls. The study group will comprise community dwelling elderly individuals over the age of 65 years who get around by themselves. After 2 years, the participants will be re-examined for their frailty and independence status, as well as their survival will be checked with the National Health Found electronic system. The aim of this project is to seek for factors determining frailty and to explore the frailty impact on the elderly people survival. Particular attention will be paid to the multidimensional frailty which is a new concept of the functional decline in the elderly. In addition, the prevalence of different modes of frailty in Polish community will be investigated. The results of this research should help to establish preventative and therapeutic strategies against frailty.

DETAILED DESCRIPTION:
Frailty is a geriatric syndrome which relies on the reduction of multisystem reserve capacity, whereas pre-frailty is a condition predisposing and preceding the frailty state. Frail people have a lower potential to respond to external stressors and various life incidents as well as they present a weak prognosis particularly in cardiovascular diseases. However, frailty is not only a set of physical deficits, but it also concerns psychological and social dimensions of human functioning. Hence, an approach to frailty should be multidimensional because such a concept more adequately reflects a functional degradation in the elderly. Frailty is usually associated with the impaired condition of circulatory system, and therefore, an identification of subclinical cardiovascular abnormalities which are associated with frailty is paramount in a context of frailty prevention and treatment. In this study, a comprehensive echocardiography will investigate cardiac function with a particular attention to features which typically change with age, like flow and diastolic parameters, as well as chambers sizes. Specifically, the impact of the impaired diastolic filling pattern on the frailty development will be thoroughly investigated. Another potential mechanism which may predispose to frailty is a dysfunction of the autonomic nervous system (ANS) - especially, its cardiac branch. ANS plays a crucial role in the response to internal or external stressors such as diseases and activities of daily living, and it plays a pivotal role in the homeostasis. Since frail people present a progressive homeostatic dysregulation, it is possible that the impairment in the cardiac ANS may maintain or accelerate the frailty process. In the present study, both tonic and reflex activities of the cardiac ANS will be explored with Finapres device (Finapres Medical Systems B.V., Amsterdam, the Netherlands) which is a gold standard for non-invasive continuous blood pressure monitoring and also allows ECG and respiratory signals recording. The study participants will also undergo routine medical examination, standard 12-lead electrocardiography, and measurements of body mass index and ankle-brachial index - the latter will reflect the degree of lower extremity arterial disease. A cognitive function and a psychological condition will be evaluated with the Mini-Mental State Examination (MMSE) and the Geriatric Depression Scale, respectively. A nutrition status will be checked with the Mini Nutritional Assessment (MNA). The Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) will be assessed with dedicated scales. A risk of fall will be judged with the questionnaire concerning the falls history and by examining a postural stability on a force plate (AccuSway, AMTI, Watertown, MA, USA). The study group will comprise community dwelling elderly individuals over the age of 65 years who get around by themselves. The exclusion criteria include: institutionalization, inability to move around, and terminal diseases with an anticipated survival of less than 1 year. After 2 and 5 years, the participants will be re-examined for their frailty and independence status, and in addition, their life status will be checked with national identification numbers by using the National Health Found registration system. Sample size calculation indicates that the minimum sample size to investigate frailty development should equal 994 subjects (1% margin of error and 95% confidence interval), however, assuming 10% loss in follow-up, the final sample size is 1093 subjects.

The primary endpoints of this study are: (i) to identify risk factors associated with multidimensional and physical frailty and pre-frailty in community dwelling elderly people over the age of 65 years; (ii) to find determinants for the development of different types of frailty in a prospective observation. The secondary endpoints are: (i) to explore the impact of various modes of frailty and other clinical factors on the elderly people mortality; (ii) to identify predictors for frailty development, disability or mortality as a composite endpoint; (iii) to explore the rate and determinants of a frailty status transition to a more robust status; (iv) to establish the prevalence of multidimensional frailty, and physical frailty and pre-frailty in elderly people in Polish community; (v) to determine a concordance/discordance between physical and multidimensional frailty.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling elderly individuals over the age of 65 years who get around by themselves.

Exclusion Criteria:

* Institutionalization
* Inability to move around
* Terminal diseases with an anticipated survival of less than 1 year.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study group will comprise community dwelling elderly individuals over the age of 65 years who get around by themselves.
Sampling Method: Probability Sample
Enrollment: 1093 (Estimated)
Dates: Start 2017-09-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Risk factors associated with multidimensional and physical frailty and pre-frailty in community dwelling elderly people over the age of 65 years. | At the study entry during the first examination.
  Risk factors associated with the existing frailty at the study entry will be identified.
Determinants for the development of different types of frailty in a prospective observation | Through the study completion, an average of 5 years.
  Determinants of frailty developing during the study period will be identified.

SECONDARY OUTCOMES:
The impact of various modes of frailty and other clinical factors on the elderly people mortality. | Through the study completion, an average of 5 years.
  Frailty impact on mortality in elderly people will be investigated.
Predictors for frailty development, disability or mortality as a composite endpoint. | Through the study completion, an average of 5 years.
  Determinants of frailty development, disability or mortality as a composite endpoint will be investigated.
The rate and determinants of a frailty status transition to a more robust status. | Through the study completion, an average of 5 years.
  The rate and determinants of the recovery from different statuses of frailty will be investigated.
The prevalence of multidimensional frailty, and physical frailty and pre-frailty in elderly people in Polish community. | Through the study completion, an average of 5 years.
  The prevalence of different types of frailty in Polish community will be investigated.
The concordance and discordance between physical and multidimensional frailty. | Through the study completion, an average of 5 years.
  The concordance and discordance between different types of frailty will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Sacha, MD, PhD, Principal Investigator — Faculty of Physical Education and Physiotherapy, Opole University of Technology
Locations (1):
- Faculty of Physical Education and Physiotherapy, Opole University of Technology, Opole, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Potentially some data will be shared for research purposes and after investigators agreement.